CLINICAL TRIAL: NCT07254052
Title: Effectiveness of a Sustained-release Ammonium Chloride Formulation in Reducing the Viral Load of Patients With COVID-19 or Influenza
Brief Title: Effectiveness of Ammonium Chloride in Reducing Viral Load
Acronym: ACTEarly
Status: Completed | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Third Department of Medicine, Sotiria General Hospital (Unknown)
Responsible Party: Principal Investigator, Nikolaos Drakoulis, MD, Professor of Clinical Pharmacology, National and Kapodistrian University of Athens
Other Study IDs: Sotiria GH 14328/17-05-2025
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: RNA Virus Infections; Viral Infection COVID-19; Influenza A and B
Keywords: ammonium chloride; influenza; SARS-CoV-2; RNA virus infections; virus clearance
MeSH Terms: conditions — RNA Virus Infections; Influenza, Human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ACF receiving participants: Participants assigned to this group received the sustained-release ammonium chloride formulation (ACF), containing 500 mg ammonium chloride and 2,000 IU vitamin D per capsule. One capsule was administered orally every 12 hours for 10 consecutive days, starting on Day 1. Both inpatients and outpatients with mild or moderate COVID-19 or seasonal influenza infection were included. The intervention aimed to evaluate the effect of ammonium chloride on viral load reduction and clinical outcomes compared to the control group. Randomization and double-blinding were maintained throughout the study.
- Control Group (VDF receiving participants): Participants assigned to this group received the control formulation consisting of sustained-release tablets containing 2,000 IU vitamin D and identical excipients, but no ammonium chloride. One capsule was administered orally every 12 hours for 10 consecutive days, starting on Day 1. Both inpatients and outpatients with mild or moderate COVID-19 or seasonal influenza infection were included. This control arm was used to compare changes in viral load dynamics and clinical outcomes against the intervention group. Randomization and double-blinding were maintained throughout the study.

SUMMARY:
This is a prospective, double-blind, randomized, comparative effectiveness pilot study evaluating the effect of a sustained-release ammonium chloride formulation (ACF) on viral load dynamics in adult patients with mild or moderate COVID-19 or seasonal influenza infection.

Eligible participants are randomly assigned in a 1:1 ratio to receive either ACF (ammonium chloride with vitamin D) or a control formulation (vitamin D only) twice daily for 10 consecutive days. The primary objective is to assess the reduction of viral load measured by RT-PCR cycle threshold (Ct) values at baseline, Day 3-5, and Day 10-12. Secondary objectives include the duration and severity of symptoms, incidence of hospitalization, oxygen supplementation, ICU admission, and mortality.

The study is conducted in both inpatient and outpatient settings at Sotiria General Hospital for Chest Diseases, Athens, Greece as well as at the outpatient clinic "En Ygeia". All viral load analyses are performed at the Department of Pharmacy, National and Kapodistrian University of Athens. A total of 32 participants were enrolled. This study aims to generate early clinical evidence regarding the antiviral effectiveness of ACF as an adjunct strategy in respiratory RNA virus infections.

DETAILED DESCRIPTION:
This is a prospective, double-blind, randomized, comparative effectiveness pilot clinical study designed to evaluate the antiviral effect of a sustained-release ammonium chloride formulation (ACF) in adult patients with mild or moderate SARS-CoV-2 or seasonal influenza infection. Respiratory viral infections remain a major global health burden, and safe, accessible adjunct therapies are needed to complement existing public health measures and vaccination strategies.

Eligible participants are adults (≥18 years) with a positive rapid test for SARS-CoV-2 or influenza A/B, recruited at the Outpatients Clinic or Emergency Department of Sotiria General Hospital for Chest Diseases and at "En Ygeia" outpatient clinic. Participants are randomized in a 1:1 ratio to receive either:

1. ACF (nutritional supplement): sustained-release ammonium chloride formulation with vitamin D, one capsule every 12 hours for 10 days
2. VDF (control): matched sustained-release placebo formulation containing only vitamin D, one capsule every 12 hours for 10 days.

Both inpatients and outpatients are included. Exclusion criteria are: age <18 years, pregnancy or lactation, denial of informed consent, known allergy to study components, organ transplantation, and frailty score ≥5. Participants may discontinue the study in cases of intolerance, non-compliance, or withdrawal of consent.

The primary endpoint is the reduction of viral load, assessed through RT-PCR cycle threshold (Ct) values obtained at baseline (Day 1), Day 3-5, and Day 10-12.

Secondary endpoints include:

* Duration and severity of symptoms for 30 days
* Incidence of hospitalization (for outpatients)
* Need for oxygen supplementation
* ICU admission
* Intubation
* Death. All RT-PCR testing for SARS-CoV-2 and influenza A/B were performed at the Department of Pharmacy, National and Kapodistrian University of Athens. The study employs standardized sampling, nucleic acid extraction, and real-time PCR quantification with certified reference materials.

Statistical analysis compared Ct values across timepoints within and between groups. Mean percentage change in Ct values was compared using appropriate parametric or non-parametric tests, with additional analyses for secondary outcomes. The final sample size was 32 patients.

This pilot trial aims to provide early clinical evidence regarding the potential antiviral effectiveness of ammonium chloride in the context of mild respiratory viral infections, contributing to the design of larger confirmatory studies.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years.
* Positive rapid test for Sars-CoV-2 19 or influenza (performed at the Outpatients Clinic or the Emergency Department).
* Informed consent.

Exclusion Criteria:

* Age < 18 years.
* Pregnancy, and/or lactation.
* Denial of Informed Consent.
* Known allergy to ammonium chloride or to any of the ACF, or VDF excipients.
* Organ transplantation.
* Frailty score ≥ 5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) with mild or moderate COVID-19 or seasonal influenza infection were recruited at the Outpatients Clinic and the Emergency Department of Sotiria General Hospital for Chest Diseases in Athens, Greece and at "En Ygeia" outpatient clinic. Both inpatients and outpatients were eligible. All participants had a laboratory-confirmed diagnosis by rapid antigen testing and were enrolled within 3-5 days of symptom onset. Patients with severe disease, organ transplantation, pregnancy, or frailty score ≥5 were excluded. A total of 32 participants completed the study procedures.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Change in viral load measured by RT-PCR Ct values | Baseline (Day 1), Day 3-5, Day 10-12
  Change in viral load was assessed through real-time PCR (RT-PCR) cycle threshold (Ct) values for SARS-CoV-2 or influenza A/B from nasopharyngeal swabs. Measurements were performed at three predefined time points (Day 1, Day 3-5, and Day 10-12). Viral load reduction was defined as an increase in Ct values over time. Samples were processed at the Department of Pharmacy, National and Kapodistrian University of Athens.

SECONDARY OUTCOMES:
Duration of symptoms | Up to Day 30 after diagnosis
  Duration of respiratory and systemic symptoms was recorded for 30 days after diagnosis. Data were collected through patient interviews and medical record review.
Hospitalization rate (outpatients only) | Up to Day 30
  Number of outpatient participants requiring hospitalization within 30 days of diagnosis.
Need for oxygen administration | Up to Day 30
  Number of participants requiring oxygen therapy during follow-up.
ICU admission | Up to Day 30
  Number of participants admitted to the ICU for respiratory deterioration.
Intubation | Up to Day 30
  Number of participants requiring endotracheal intubation.
Mortality | Up to Day 30
  Number of deaths from any cause during the 30-day follow-up period.

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - En Ygeia Clinic, Athens
  - Sotiria General Hospital, Athens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeichhardt H, Wetz K, Willingmann P, Habermehl KO. Entry of poliovirus type 1 and Mouse Elberfeld (ME) virus into HEp-2 cells: receptor-mediated endocytosis and endosomal or lysosomal uncoating. J Gen Virol. 1985 Mar;66 ( Pt 3):483-92. doi: 10.1099/0022-1317-66-3-483. PMID 2857762
- [Background] Yoshimura A, Ohnishi S. Uncoating of influenza virus in endosomes. J Virol. 1984 Aug;51(2):497-504. doi: 10.1128/JVI.51.2.497-504.1984. PMID 6431119
- [Background] Superti F, Seganti L, Orsi N, Divizia M, Gabrieli R, Pana A. The effect of lipophilic amines on the growth of hepatitis A virus in Frp/3 cells. Arch Virol. 1987;96(3-4):289-96. doi: 10.1007/BF01320970. PMID 2821967
- [Background] Silva PJS, Sagastizabal C, Nonato LG, Struchiner CJ, Pereira T. Optimized delay of the second COVID-19 vaccine dose reduces ICU admissions. Proc Natl Acad Sci U S A. 2021 Aug 31;118(35):e2104640118. doi: 10.1073/pnas.2104640118. PMID 34408076
- [Background] Shrestha LB, Foster C, Rawlinson W, Tedla N, Bull RA. Evolution of the SARS-CoV-2 omicron variants BA.1 to BA.5: Implications for immune escape and transmission. Rev Med Virol. 2022 Sep;32(5):e2381. doi: 10.1002/rmv.2381. Epub 2022 Jul 20. PMID 35856385
- [Background] Shi T, Denouel A, Tietjen AK, Campbell I, Moran E, Li X, Campbell H, Demont C, Nyawanda BO, Chu HY, Stoszek SK, Krishnan A, Openshaw P, Falsey AR, Nair H; RESCEU Investigators. Global Disease Burden Estimates of Respiratory Syncytial Virus-Associated Acute Respiratory Infection in Older Adults in 2015: A Systematic Review and Meta-Analysis. J Infect Dis. 2020 Oct 7;222(Suppl 7):S577-S583. doi: 10.1093/infdis/jiz059. PMID 30880339
- [Background] Shang C, Zhuang X, Zhang H, Li Y, Zhu Y, Lu J, Ge C, Cong J, Li T, Tian M, Jin N, Li X. Inhibitors of endosomal acidification suppress SARS-CoV-2 replication and relieve viral pneumonia in hACE2 transgenic mice. Virol J. 2021 Feb 27;18(1):46. doi: 10.1186/s12985-021-01515-1. PMID 33639976
- [Background] Prabhakara C, Godbole R, Sil P, Jahnavi S, Gulzar SE, van Zanten TS, Sheth D, Subhash N, Chandra A, Shivaraj A, Panikulam P, U I, Nuthakki VK, Puthiyapurayil TP, Ahmed R, Najar AH, Lingamallu SM, Das S, Mahajan B, Vemula P, Bharate SB, Singh PP, Vishwakarma R, Guha A, Sundaramurthy V, Mayor S. Strategies to target SARS-CoV-2 entry and infection using dual mechanisms of inhibition by acidification inhibitors. PLoS Pathog. 2021 Jul 12;17(7):e1009706. doi: 10.1371/journal.ppat.1009706. eCollection 2021 Jul. PMID 34252168
- [Background] Pifarre I Arolas H, Acosta E, Lopez-Casasnovas G, Lo A, Nicodemo C, Riffe T, Myrskyla M. Years of life lost to COVID-19 in 81 countries. Sci Rep. 2021 Feb 18;11(1):3504. doi: 10.1038/s41598-021-83040-3. PMID 33603008
- [Background] Nguyen NN, Houhamdi L, Hoang VT, Stoupan D, Fournier PE, Raoult D, Colson P, Gautret P. High rate of reinfection with the SARS-CoV-2 Omicron variant. J Infect. 2022 Aug;85(2):174-211. doi: 10.1016/j.jinf.2022.04.034. Epub 2022 Apr 23. No abstract available. PMID 35472367
- [Background] Mizzen L, Hilton A, Cheley S, Anderson R. Attenuation of murine coronavirus infection by ammonium chloride. Virology. 1985 Apr 30;142(2):378-88. doi: 10.1016/0042-6822(85)90345-9. PMID 2997991
- [Background] Maltezou HC, Raftopoulos V, Vorou R, Papadima K, Mellou K, Spanakis N, Kossyvakis A, Gioula G, Exindari M, Froukala E, Martinez-Gonzalez B, Panayiotakopoulos G, Papa A, Mentis A, Tsakris A. Association Between Upper Respiratory Tract Viral Load, Comorbidities, Disease Severity, and Outcome of Patients With SARS-CoV-2 Infection. J Infect Dis. 2021 Apr 8;223(7):1132-1138. doi: 10.1093/infdis/jiaa804. PMID 33388780
- [Background] Maltezou HC, Papanikolopoulou A, Vassiliu S, Theodoridou K, Nikolopoulou G, Sipsas NV. COVID-19 and Respiratory Virus Co-Infections: A Systematic Review of the Literature. Viruses. 2023 Mar 28;15(4):865. doi: 10.3390/v15040865. PMID 37112844
- [Background] Maltezou HC, Papadima K, Gkolfinopoulou K, Ferentinos G, Mouratidou E, Andreopoulou A, Pavli A, Magaziotou I, Georgakopoulou T, Mellou K, Vorou R, Antoniadou A, Stathakarou A, Chrysochoou A, Gogos C, Karaiskou A, Kotanidou A, Koutsoukou A, Marangos M, Mentis A, Metallidis S, Papa A, Pefanis A, Tsakris A, Sipsas NV. Coronavirus disease 2019 pandemic in Greece, February 26 - May 3, 2020: The first wave. Travel Med Infect Dis. 2021 May-Jun;41:102051. doi: 10.1016/j.tmaid.2021.102051. Epub 2021 Apr 2. No abstract available. PMID 33819570
- [Background] Maltezou HC, Krumbholz B, Mavrouli M, Tseroni M, Gamaletsou MN, Botsa E, Anastassopoulou C, Gikas A, Fournarakou E, Kavieri M, Koureli A, Mandilara D, Marinopoulou A, Theodorikakou A, Tsiahris P, Zarzali A, Pournaras S, Lourida A, Elefsiniotis I, Vrioni G, Sipsas NV, Tsakris A. A study of the evolution of the third COVID-19 pandemic wave in the Athens metropolitan area, Greece, through two cross-sectional seroepidemiological surveys: March, June 2021. J Med Virol. 2022 Apr;94(4):1465-1472. doi: 10.1002/jmv.27465. Epub 2021 Dec 4. PMID 34812522
- [Background] Li Y, Wang X, Blau DM, Caballero MT, Feikin DR, Gill CJ, Madhi SA, Omer SB, Simoes EAF, Campbell H, Pariente AB, Bardach D, Bassat Q, Casalegno JS, Chakhunashvili G, Crawford N, Danilenko D, Do LAH, Echavarria M, Gentile A, Gordon A, Heikkinen T, Huang QS, Jullien S, Krishnan A, Lopez EL, Markic J, Mira-Iglesias A, Moore HC, Moyes J, Mwananyanda L, Nokes DJ, Noordeen F, Obodai E, Palani N, Romero C, Salimi V, Satav A, Seo E, Shchomak Z, Singleton R, Stolyarov K, Stoszek SK, von Gottberg A, Wurzel D, Yoshida LM, Yung CF, Zar HJ; Respiratory Virus Global Epidemiology Network; Nair H; RESCEU investigators. Global, regional, and national disease burden estimates of acute lower respiratory infections due to respiratory syncytial virus in children younger than 5 years in 2019: a systematic analysis. Lancet. 2022 May 28;399(10340):2047-2064. doi: 10.1016/S0140-6736(22)00478-0. Epub 2022 May 19. PMID 35598608
- [Background] Helenius A, Marsh M, White J. Inhibition of Semliki forest virus penetration by lysosomotropic weak bases. J Gen Virol. 1982 Jan;58 Pt 1:47-61. doi: 10.1099/0022-1317-58-1-47. PMID 7142969
- [Background] Grange Z, Buelo A, Sullivan C, Moore E, Agrawal U, Boukhari K, McLaughlan I, Stockton D, McCowan C, Robertson C, Sheikh A, Murray JLK. Characteristics and risk of COVID-19-related death in fully vaccinated people in Scotland. Lancet. 2021 Nov 13;398(10313):1799-1800. doi: 10.1016/S0140-6736(21)02316-3. Epub 2021 Oct 28. No abstract available. PMID 34756204
- [Background] Georgakopoulou VE, Vlachogiannis NI, Basoulis D, Eliadi I, Georgiopoulos G, Karamanakos G, Makrodimitri S, Samara S, Triantafyllou M, Voutsinas PM, Ntziora F, Psichogiou M, Samarkos M, Sfikakis PP, Sipsas NV. A Simple Prognostic Score for Critical COVID-19 Derived from Patients without Comorbidities Performs Well in Unselected Patients. J Clin Med. 2022 Mar 25;11(7):1810. doi: 10.3390/jcm11071810. PMID 35407418
- [Background] Fournier PE, Houhamdi L, Colson P, Cortaredona S, Delorme L, Cassagne C, Lagier JC, Chaudet H, Tissot-Dupont H, Giraud-Gatineau A, Fenollar F, Million M, Raoult D. SARS-CoV-2 Vaccination and Protection Against Clinical Disease: A Retrospective Study, Bouches-du-Rhone District, Southern France, 2021. Front Microbiol. 2022 Jan 18;12:796807. doi: 10.3389/fmicb.2021.796807. eCollection 2021. PMID 35116013
- [Background] Faust JS, Chen AJ, Nguemeni Tiako MJ, Du C, Li SX, Krumholz HM, Barnett ML. Leading Causes of Death Among Adults Aged 25 to 44 Years by Race and Ethnicity in Texas During the COVID-19 Pandemic, March to December 2020. JAMA Intern Med. 2022 Jan 1;182(1):87-90. doi: 10.1001/jamainternmed.2021.6734. PMID 34807250
- [Background] Qu P, Faraone J, Evans JP, Zou X, Zheng YM, Carlin C, Bednash JS, Lozanski G, Mallampalli RK, Saif LJ, Oltz EM, Mohler PJ, Gumina RJ, Liu SL. Neutralization of the SARS-CoV-2 Omicron BA.4/5 and BA.2.12.1 Subvariants. N Engl J Med. 2022 Jun 30;386(26):2526-2528. doi: 10.1056/NEJMc2206725. Epub 2022 Jun 15. No abstract available. PMID 35704428
- [Background] Siami Z, Aghajanian S, Mansouri S, Mokhames Z, Pakzad R, Kabir K, Norouzi M, Soleimani A, Hedayat Yaghoobi M, Shadabi S, Tajbakhsh R, Kargar Kheirabad A, Mozhgani SH. Effect of Ammonium Chloride in addition to standard of care in outpatients and hospitalized COVID-19 patients: A randomized clinical trial. Int J Infect Dis. 2021 Jul;108:306-308. doi: 10.1016/j.ijid.2021.04.043. Epub 2021 Apr 18. PMID 33878462
- [Background] Hidvegi M, Nichelatti M. Bacillus Calmette-Guerin vaccination Policy and Consumption of Ammonium Chloride-Enriched Confectioneries May Be Factors Reducing COVID-19 Death Rates in Europe. Isr Med Assoc J. 2020 Aug;22(8):501-504. PMID 33236583
- [Background] Di Trani L, Savarino A, Campitelli L, Norelli S, Puzelli S, D'Ostilio D, Vignolo E, Donatelli I, Cassone A. Different pH requirements are associated with divergent inhibitory effects of chloroquine on human and avian influenza A viruses. Virol J. 2007 May 3;4:39. doi: 10.1186/1743-422X-4-39. PMID 17477867
- [Background] Chemaitelly H, Ayoub HH, AlMukdad S, Coyle P, Tang P, Yassine HM, Al-Khatib HA, Smatti MK, Hasan MR, Al-Kanaani Z, Al-Kuwari E, Jeremijenko A, Kaleeckal AH, Latif AN, Shaik RM, Abdul-Rahim HF, Nasrallah GK, Al-Kuwari MG, Butt AA, Al-Romaihi HE, Al-Thani MH, Al-Khal A, Bertollini R, Abu-Raddad LJ. Duration of mRNA vaccine protection against SARS-CoV-2 Omicron BA.1 and BA.2 subvariants in Qatar. Nat Commun. 2022 Jun 2;13(1):3082. doi: 10.1038/s41467-022-30895-3. PMID 35654888
- [Background] Bar-On YM, Goldberg Y, Mandel M, Bodenheimer O, Amir O, Freedman L, Alroy-Preis S, Ash N, Huppert A, Milo R. Protection by a Fourth Dose of BNT162b2 against Omicron in Israel. N Engl J Med. 2022 May 5;386(18):1712-1720. doi: 10.1056/NEJMoa2201570. Epub 2022 Apr 5. PMID 35381126
- [Background] Cicero AFG, Fogacci F, Borghi C. Vitamin D Supplementation and COVID-19 Outcomes: Mounting Evidence and Fewer Doubts. Nutrients. 2022 Aug 31;14(17):3584. doi: 10.3390/nu14173584. PMID 36079842